CLINICAL TRIAL: NCT01751113
Title: A Randomised, Double-blind, Double Dummy, 3 Way Cross-over Study Evaluating the Effects of ADOAIR 50/250mcg Twice Daily Plus Tiotropium Bromide 18mcg Once Daily Compared With the Individual Treatments (Tiotropium Bromide 18mcg Alone and ADOAIR 50/250mcg Alone) in the Treatment of Japanese Subjects With COPD
Brief Title: A 3 Way Cross-over Study Evaluating the Effects of ADOAIR Twice Daily Plus Tiotropium Bromide Once Daily Compared With the Individual Treatments of Japanese Subjects
Acronym: SCO116572
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116572
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; Tiotropium Bromide; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- fluticasone propionate/salmeterol (Active Comparator): 250mcg fluticasone + 50 mcg salmeterol, twice daily 4 week treatment in each treatment sequence (crossover design)
  Interventions: Drug: fluticasone propionate/salmeterol
- tiotropium bromide (Active Comparator): 18 mcg tiotropium bromide, once daily 4 week treatment in each treatment sequence (crossover design)
  Interventions: Drug: tiotropium bromide
- fluticasone propionate/salmeterol plus tiotropium bromide (Active Comparator): 250mcg fluticasone + 50 mcg salmeterol, twice daily plus 18 mcg tiotropium bromide, once daily 4 week treatment in each treatment sequence (crossover design)
  Interventions: Drug: fluticasone propionate/salmeterol plus tiotropium bromide

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol — 250mcg fluticasone + 50 mcg salmeterol, twice daily 4 week treatment in each treatment sequence (crossover design)
  Other Names: ADOAIR is a registered trade mark of the GlaxoSmithKlline group of companies.
  Arms: fluticasone propionate/salmeterol
Drug: tiotropium bromide — 18 mcg tiotropium bromide, once daily 4 week treatment in each treatment sequence (crossover design)
  Arms: tiotropium bromide
Drug: fluticasone propionate/salmeterol plus tiotropium bromide — 250mcg fluticasone + 50 mcg salmeterol, twice daily plus 18 mcg tiotropium bromide, once daily 4 week treatment in each treatment sequence (crossover design)
  Other Names: ADOAIR is a registered trade mark of the GlaxoSmithKlline group of companies.
  Arms: fluticasone propionate/salmeterol plus tiotropium bromide

SUMMARY:
The purpose of this study is to evaluate the effects on lung function of a combination of ADOAIR 50/250mcg twice daily plus tiotropium bromide 18mcg once daily compared with the individual treatments (tiotropium bromide 18mcg once daily alone and ADOAIR 50/250mcg twice daily alone) in Japanese subjects with COPD. The study will utilize a three-way cross-over design with a 2-week wash-out period between each 4-week consecutive treatment period. The aim is to support the rationale for "triple combination" therapy by demonstrating that treatment with both ADOAIR and tiotropium can potentially produce improved, clinically relevant effects compared with either treatment alone.

This study will utilize a range of lung function measures in order to fully assess the benefits of triple therapy. The primary endpoint will be based on airways conductance measured using plethysmography (sGaw measured over 4hours post dose (AUC 0-4hr) on Day 28). Secondary endpoints will include lung function measures based on plethysmography and spirometry. The lung function measures will be supported by measurement of the use of relief salbutamol .

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 40 - 80 years inclusive
* Has an established clinical history of COPD (defined as per the GOLD definition)
* A signed and dated written informed consent is obtained from the subject prior to study participation
* The subject has a post-bronchodilator FEV1 of >=30% to =<75% of predicted normal at Visit 1
* The subject has a post-bronchodilator FEV1/ FVC ratio <70% at Visit 1
* The subject achieves a score of 1 on the Modified Medical Research Council (mMRC) Dyspnoea Scale at Visit 1
* The subject is a current or ex-smoker with a smoking history of > 10 pack-years (10 pack years is defined as 20 cigarettes per day for 10 years, or 10 cigarettes (or equivalent if subject smoked cigars or a pipe) per day for 20 years). Ex-smokers are required to have stopped smoking for at least 6 months prior to visit 1. Ex-smokers who stopped smoking less than 6 months ago will be defined as current smokers.
* QTc <450 msec at Visit 1; or for patients with Bundle Branch Block QTc should be <480 msec.

(QTc(F) <450msec, or <480 in subjects with right bundle branch block, should be confirmed by the mean of three readings or one reading)

* ALT < 2xULN and bilirubin/ALP < 1.5xULN (>35% direct bilirubin)
* A female is eligible to enter this study if she is: i)of non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal), ii)of child-bearing potential, but has a negative urinary pregnancy test at screening and agrees to take contraceptive precautions (including abstinence) which are adequate to prevent pregnancy during the study or iii)not a nursing mother

Exclusion Criteria:

* Has had a COPD exacerbation within the 4 weeks prior to Visit 1
* Had any changes in COPD medication in the 4 weeks prior to Visit 1
* Has plan to change the dosage of Xanthines or to stop receiving it during the study
* Has a current medical diagnosis of asthma
* Has a medical diagnosis of narrow-angle glaucoma, prostatic hyperplasia or bladder neck obstruction that in the opinion of the investigator should prevent them from entering the study Note: As with other anticholinergic drugs, subjects with narrow-angle glaucoma, prostatic hyperplasia or bladder neck obstruction should only be entered into the study at the Investigator's discretion
* Has known respiratory disorders other than COPD (e.g. lung cancer, sarcoidosis, tuberculosis or lung fibrosis)
* Has undergone lung surgery e.g., lung transplant and/or lung volume reduction
* Is currently receiving pulmonary rehabilitation
* Had a chest X-ray indicating diagnosis other than COPD that might interfere with the study (chest X-ray to be taken at entry, if subject has not had one or CT image taken within 3 months of Visit 1)
* Requires regular (daily) or long term oxygen therapy (LTOT). (LTOT is defined as . 12 hours oxygen use per day)
* Requires regular treatment with oral, parenteral, or depot corticosteroids or has received 2 or more periods of oral corticosteroids for COPD exacerbation in the last 6 months
* Received oral, parenteral, or depot corticosteroids in the 4 weeks prior to Visit 1
* Received antibiotic therapy for either a lower respiratory tract infection or for COPD exacerbation within the 4 weeks prior to Visit 1
* Has been hospitalized for a COPD exacerbation in the last year
* Receiving non-selective β-blockers (except eye drops)
* Has serious, uncontrolled disease likely to interfere with the study (e.g. Left Ventricular failure, anaemia, renal or hepatic disease or serious psychological disorders)
* Received any other investigational drugs within 4 weeks (or 5 half lives) prior to Visit 1
* Has, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse
* Has a known or suspected hypersensitivity to β2-agonists, inhaled steroids, anticholinergic treatments or any components of the formulations (e.g. lactose or milk protein)
* Has previously been enrolled and randomized to this study
* Are not considered able to tolerate three 2-weeks wash-out periods according to the study schedule with all COPD medications removed apart from rescue use of SALBUTAMOL via MDI (inhaled PRN use).
* Is not eligible to participate this study in the opinion of the investigator/subinvestigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Japan (3):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 116572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 53 Japanese participants with moderate or severe chronic obstructive pulmonary disease (COPD) entered the run-in period.
Pre-assignment Details: Participants, who met eligibility criteria, completed a 2-week Run-in Period prior to being randomized to 1 of 6 treatment sequences. The treatment phase was comprised of three 4 week treatment periods, each separated by a 2-week washout period.
Groups:
- Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg: Participants received salmeterol xinafoate/fluticasone propionate (Ado) 50/250 micrograms (µg) twice daily (BID) (morning and evening) plus tiotropium bromide (Tio) 18 µg once daily (QD) (morning), Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening), and Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning) in Treatment Periods 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via a HandiHaler inhaler. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg: Participants received Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening), Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning), and Ado 50/250 µg BID plus Tio 18 µg QD (morning) in Treatment Periods 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via a HandiHaler inhaler. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg: Participants received Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning), Ado 50/250 µg BID plus Tio 18 µg QD (morning), and Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening) in Treatment Period 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via HandiHaler inhaler. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg: Participants received Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning), Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening), and Ado 50/250 µg BID plus Tio 18 µg QD (morning) in Treatment Period 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via a HandiHaler inhaler. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg: Participants received Ado 50/250 µg BID plus Tio 18 µg QD (morning), Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning) and Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening) in Treatment Period 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via a HandiHaler inhaler. Participants were provided with salbutamol inhaler to be used as relief medication throughout the study.
- Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg: Participants received Tio 18 µg QD (morning) plus Ado matching placebo BID (morning and evening), Ado 50/250 µg BID plus Tio 18 µg QD (morning), and Ado 50/250 µg BID (morning and evening) plus Tio matching placebo QD (morning) in Treatment Period 1, 2, and 3, respectively. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Ado 50/250 µg and its matching placebo were administered via a dry powder inhaler and Tio 18 µg and its matching placebo were administered via a HandiHaler inhaler. Participants were provided with salbutamol inhaler to be used as relief medication throughout the study.
Period: Treatment Period 1 (4 Weeks)
Arm/Group | Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg | Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg | Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg | Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg | Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg | Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg
Started | 8 | 8 | 9 | 9 | 9 | 10
Completed | 8 | 8 | 9 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Period: Washout Period 1 (2 Weeks)
Arm/Group | Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg | Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg | Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg | Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg | Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg | Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg
Started | 8 | 8 | 9 | 8 | 8 | 10
Completed | 8 | 8 | 9 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (4 Weeks)
Arm/Group | Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg | Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg | Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg | Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg | Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg | Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg
Started | 8 | 8 | 9 | 8 | 8 | 10
Completed | 8 | 8 | 9 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (2 Weeks)
Arm/Group | Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg | Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg | Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg | Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg | Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg | Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg
Started | 8 | 8 | 9 | 8 | 8 | 10
Completed | 8 | 8 | 9 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (4 Weeks)
Arm/Group | Sequence 1: Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg | Sequence 2: Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg | Sequence 3: Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg | Sequence 4: Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg | Sequence 5: Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg | Sequence 6: Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg
Started | 8 | 8 | 9 | 8 | 8 | 10
Completed | 8 | 8 | 9 | 8 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg: All participants received one of the following 3 treatments in one of three 4-week treatment periods separated by a 2-week washout period:Ado 50/250 µg BID (morning and evening) + Tio 18 µg QD (morning), Ado 50/250 µg BID (morning and evening) + Tio matching placebo QD (morning), and Tio 18 µg QD (morning) + Ado matching placebo BID (morning and evening). Participants were randomized to one of the 6 following treatment sequences: (1) Ado 50/250 µg+Tio 18 µg, Tio 18 µg, Ado 50/250 µg (2) Tio 18 µg, Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg (3) Ado 50/250 µg, Ado 50/250 µg+Tio 18 µg, Tio 18 µg (4) Ado 50/250 µg, Tio 18 µg, Ado 50/250 µg+Tio 18 µg (5) Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg (6) Tio 18 µg, Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg. Ado 50/250 µg and its matching placebo were administered via DISKUS inhaler and Tio 18 µg and its matching placebo were administered via HandiHaler inhaler. Participants used salbutamol inhaler as relief medication throughout the study.
Arm/Group | Ado 50/250 µg+Tio 18 µg, Ado 50/250 µg, Tio 18 µg
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 52
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 53

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve Calculated From 0 to 4 Hours (AUC[0-4hr]) Specific Conductance (sGaw) After the Morning Dose of Study Medication at Day 28 of Each Treatment Period
Description: sGaw is a measure of airways conductance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Plethysmography was performed to assess sGaw. The AUC was determined by using the trapezoidal rule and then dividing by the relevant time interval. A natural logarithmic transformation was applied and the data was analyzed by a mixed model including treatment, period and Baseline sGaw fitted as fixed effects and participants fitted as a random effect. Treatment ratios of all statistical comparisons were calculated by taking the anti-log of the difference between the Least Square (LS) means.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants who received at least one dose of study medication and completed at least two treatment periods and also had a Baseline and at least one on treatment sGaw assessment measure.
Measure: Geometric Mean (Standard Error); unit: 1/kilopascal*second (1/kPa*s)
Groups:
- Ado 50/250 µg BID+Tio 18 µg QD: Participants received Ado 50/250 µg BID (morning and evening) via a dry powder inhaler plus Tio 18 µg QD (morning) via a HandiHaler inhaler, in one of the three treatment periods. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Tio 18 µg QD: Participants received Tio 18 µg QD (morning) via a HandiHaler inhaler plus Ado matching placebo BID (morning and evening) via dry powder inhaler, in one of the three treatment periods. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
- Ado 50/250 µg BID: Participants received Ado 50/250 µg BID (morning and evening) via a dry powder inhaler plus Tio matching placebo QD (morning) via a HandiHaler inhaler, in one of the three treatment periods. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
1/kilopascal*second (1/kPa*s) | 0.854 (0.0183) | 0.737 (0.0183) | 0.663 (0.0182)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; AUC ratio = 1.158, 95% CI 2-sided [1.100 to 1.219]
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; AUC ratio = 1.288, 95% CI 2-sided [1.224 to 1.355]

2. Secondary Outcome: AUC (0-4hr) Specific Airway Resistance (sRaw) After the Morning Dose of Each Study Medication at Day 28 of Each Treatment Period
Description: sRaw is a measure of airways resistance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Plethysmography was performed to assess sRaw. The AUC was determined by using the trapezoidal rule and then dividing by the relevant time interval. A natural logarithmic transformation was applied and the data was analyzed by a mixed model including treatment, period and Baseline sRaw fitted as fixed effects and participants fitted as a random effect. Treatment ratios of all statistical comparisons were calculated by taking the anti-log of the difference between the LS means.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Geometric Mean (Standard Error); unit: kPa*s
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
kPa*s | 1.181 (0.0188) | 1.380 (0.0189) | 1.525 (0.0188)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; AUC ratio = 0.856, 95% CI 2-sided [0.812 to 0.902]
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; AUC ratio = 0.774, 95% CI 2-sided [0.735 to 0.816]

3. Secondary Outcome: Post-dose sGaw at 30, 75, 120 and 240 Minutes Post Dose at Day 28 of Each Treatment Period
Description: sGaw is a measure of airways conductance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Plethysmography was performed to assess sGaws. A natural logarithmic transformation was applied and the data was analyzed by a mixed model including treatment, time, period, a treatment by time interaction and Baseline sGaw fitted as fixed effects and participant fitted as a random effect.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Geometric Mean (Standard Error); unit: 1/kPa*s
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
1/kPa*s
  30 min | 0.833 (0.0241) | 0.705 (0.0241) | 0.639 (0.0240)
  75 min | 0.873 (0.0241) | 0.743 (0.0241) | 0.652 (0.0240)
  120 min | 0.885 (0.0241) | 0.769 (0.0241) | 0.680 (0.0240)
  240 min | 0.855 (0.0241) | 0.750 (0.0241) | 0.690 (0.0240)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.181, 95% CI 2-sided [1.104 to 1.263] — Statistical data for 30 minutes
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.303, 95% CI 2-sided [1.219 to 1.393] — Statistical data for 30 minutes
Statistical Analysis 3: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.175, 95% CI 2-sided [1.099 to 1.257] — Statistical data for 75 minutes
Statistical Analysis 4: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.340, 95% CI 2-sided [1.253 to 1.432] — Statistical data for 75 minutes
Statistical Analysis 5: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.151, 95% CI 2-sided [1.076 to 1.231] — Statistical data for 120 minutes
Statistical Analysis 6: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.301, 95% CI 2-sided [1.217 to 1.391] — Statistical data for 120 minutes
Statistical Analysis 7: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.141, 95% CI 2-sided [1.067 to 1.220] — Statistical data for 240 minutes
Statistical Analysis 8: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.239, 95% CI 2-sided [1.159 to 1.325] — Statistical data for 240 minutes

4. Secondary Outcome: Post-dose sRaw at 30, 75, 120 and 240 Minutes Post Dose at Day 28 of Each Treatment Period
Description: sRaw is a measure of airways resistance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Plethysmography was performed to assess sRaw. A natural logarithmic transformation was applied and the data was analysed by a mixed model including treatment, time, period, a treatment by time interaction and Baseline sRaw fitted as fixed effects and participant fitted as a random effect.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Geometric Mean (Standard Error); unit: kPa*s
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
kPa*s
  30 min | 1.201 (0.0240) | 1.419 (0.0240) | 1.567 (0.0240)
  75 min | 1.146 (0.0240) | 1.348 (0.0240) | 1.535 (0.0240)
  120 min | 1.129 (0.0240) | 1.300 (0.0240) | 1.468 (0.0240)
  240 min | 1.170 (0.0240) | 1.334 (0.0240) | 1.446 (0.0240)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.846, 95% CI 2-sided [0.792 to 0.905] — Statistical data for 30 minutes
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.767, 95% CI 2-sided [0.717 to 0.819] — Statistical data for 30 minutes
Statistical Analysis 3: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.850, 95% CI 2-sided [0.795 to 0.909] — Statistical data for 75 minutes
Statistical Analysis 4: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.746, 95% CI 2-sided [0.698 to 0.798] — Statistical data for 75 minutes
Statistical Analysis 5: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.868, 95% CI 2-sided [0.812 to 0.928] — Statistical data for 120 minutes
Statistical Analysis 6: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.769, 95% CI 2-sided [0.719 to 0.822] — Statistical data for 120 minutes
Statistical Analysis 7: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.877, 95% CI 2-sided [0.820 to 0.938] — Statistical data for 240 minutes
Statistical Analysis 8: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.809, 95% CI 2-sided [0.757 to 0.865] — Statistical data for 240 minutes

5. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1), Forced Vital Capacity (FVC), Inspiratory Capacity (IC), RV, TLC, and TGV at Each Clinic Visit Prior to the Morning Dose and Before the Use of Rescue Medication at Day 28 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration. FEV1 and FVC data was obtained by spirometry measurements. IC is defined as the maximum amount of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Total lung capacity (TLC) is the maximum volume to which the lungs can be expanded with the greatest possible inspiratory effort; it is equal to the vital capacity (VC) plus the residual volume (RV). RV is defined as the volume of air remaining in the lungs. after a maximal exhalation. Thoracic gas volume at functional residual capacity (TGV) is defined as the volume of intrathoracic gas at the time the airway is occluded for the plethysmographic measurement at the end of a normal expiration. Trough values were the values taken pre-dose.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
Liters (L)
  FEV1 | 1.823 (0.0147) | 1.666 (0.0147) | 1.706 (0.0147)
  FVC | 3.575 (0.0182) | 3.493 (0.0182) | 3.439 (0.0182)
  IC | 2.460 (0.0177) | 2.406 (0.0179) | 2.395 (0.0174)
  RV | 3.021 (0.0282) | 3.129 (0.0286) | 3.123 (0.0278)
  TLC | 6.511 (0.0189) | 6.524 (0.0191) | 6.525 (0.0186)
  TGV | 4.053 (0.0206) | 4.118 (0.0210) | 4.129 (0.0204)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean difference of FEV1 = 0.157, 95% CI 2-sided [0.116 to 0.198] — Statistical data for FEV1
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean difference of FEV1 = 0.118, 95% CI 2-sided [0.077 to 0.159] — Statistical data for FEV1
Statistical Analysis 3: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; Mean difference of FVC = 0.082, 95% CI 2-sided [0.031 to 0.133] — Statistical data for FVC
Statistical Analysis 4: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean difference of FVC = 0.135, 95% CI 2-sided [0.084 to 0.186] — Statistical data for FVC
Statistical Analysis 5: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.035, Mixed Models Analysis; Mean difference of IC = 0.054, 95% CI 2-sided [0.004 to 0.104] — Statistical data for IC
Statistical Analysis 6: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; Mean difference of IC = 0.064, 95% CI 2-sided [0.015 to 0.114] — Statistical data for IC
Statistical Analysis 7: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; Mean difference of RV = -0.107, 95% CI 2-sided [-0.187 to -0.028] — Statistical data for RV
Statistical Analysis 8: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Mean difference of RV = -0.102, 95% CI 2-sided [-0.180 to -0.023] — Statistical data for RV
Statistical Analysis 9: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.632, Mixed Models Analysis; Mean difference of TLC = -0.013, 95% CI 2-sided [-0.066 to 0.040] — Statistical data for TLC
Statistical Analysis 10: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.596, Mixed Models Analysis; Mean difference of TLC = -0.014, 95% CI 2-sided [-0.067 to 0.038] — Statistical data for TLC
Statistical Analysis 11: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; Mean difference of TGV = -0.065, 95% CI 2-sided [-0.123 to -0.007] — Statistical data for TGV
Statistical Analysis 12: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; Mean difference of TGV = -0.075, 95% CI 2-sided [-0.133 to -0.018] — Statistical data for TGV

6. Secondary Outcome: Trough FEV1/FVC Ratio, at Each Clinic Visit Prior to the Morning Dose and Before the Use of Rescue Medication at Day 28 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration. FEV1 and FVC data was obtained by spirometry measurements. Trough values were the values taken pre-dose.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Ratio of FEV1/FVC
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
Ratio of FEV1/FVC | 0.513 (0.0032) | 0.481 (0.0032) | 0.496 (0.0032)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; FEV1/FVC ratio = 0.032, 95% CI 2-sided [0.023 to 0.041] — Statistical data for FEV1/FVC ratio
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; FEV1/FVC ratio = 0.017, 95% CI 2-sided [0.008 to 0.026] — Statistical data for FEV1/FVC ratio

7. Secondary Outcome: Trough sRaw Measured at Each Clinic Visit Prior to the Morning Dose and Before the Use of Rescue Medication at Day 28 of Each Treatment Period
Description: sRaw is a measure of airways resistance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Trough values were the values taken pre-dose.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Geometric Mean (Standard Error); unit: kPa*s
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
kPa*s | 1.391 (0.0288) | 1.666 (0.0286) | 1.732 (0.0284)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.835, 95% CI 2-sided [0.770 to 0.905]
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 0.803, 95% CI 2-sided [0.741 to 0.869]

8. Secondary Outcome: Trough sGaw Measured at Each Clinic Visit Prior to the Morning Dose and Before the Use of Rescue Medication at Day 28 of Each Treatment Period
Description: sGaw is a measure of airways conductance and is intimately related to the diameter of the airways and consequently the level of bronchodilation. Trough values were the values taken pre-dose.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Geometric Mean (Standard Error); unit: 1/kPa*s
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
1/kPa*s | 0.720 (0.0287) | 0.600 (0.0285) | 0.577 (0.0284)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.200, 95% CI 2-sided [1.108 to 1.301]
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; specific airway conductance ratio = 1.249, 95% CI 2-sided [1.153 to 1.352]

9. Secondary Outcome: Post-dose FEV1, FVC, IC, RV, TLC and TGV (Measured at Trough) at Day 28 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration. FEV1 and FVC data was obtained by spirometry measurements. IC is defined as the maximum amount of air that can be inhaled into the lungs from the normal resting position after breathing out normally. Total lung capacity (TLC) is the maximum volume to which the lungs can be expanded with the greatest possible inspiratory effort; it is equal to the vital capacity (VC) plus the RV. RV is defined as the volume of air remaining in the lungs after a maximal exhalation. Thoracic gas volume at functional residual capacity (TGV) is defined as the volume of intrathoracic gas at the time the airway is occluded for the plethysmographic measurement at the end of a normal expiration.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
Liters (L)
  FEV1 | 1.766 (0.0269) | 1.605 (0.0269) | 1.664 (0.0269)
  FVC | 3.535 (0.0403) | 3.430 (0.0403) | 3.387 (0.0403)
  IC | 2.344 (0.0415) | 2.351 (0.0414) | 2.351 (0.0405)
  RV | 3.045 (0.0543) | 3.275 (0.0542) | 3.234 (0.0533)
  TLC | 6.487 (0.0395) | 6.588 (0.0394) | 6.592 (0.0386)
  TGV | 4.147 (0.0414) | 4.239 (0.0414) | 4.238 (0.0405)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean difference of FEV1 = 0.161, 95% CI 2-sided [0.086 to 0.236] — Statistical data for FEV1
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Mean difference of FEV1 = 0.103, 95% CI 2-sided [0.028 to 0.178] — Statistical data for FEV1
Statistical Analysis 3: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis; Mean difference of FVC = 0.104, 95% CI 2-sided [0.000 to 0.209] — Statistical data for FVC
Statistical Analysis 4: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Mean difference of FVC = 0.148, 95% CI 2-sided [0.043 to 0.253] — Statistical data for FVC
Statistical Analysis 5: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.890, Mixed Models Analysis; Mean difference of IC = -0.008, 95% CI 2-sided [-0.120 to 0.104] — Statistical data for IC
Statistical Analysis 6: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.890, Mixed Models Analysis; Mean difference of IC = -0.008, 95% CI 2-sided [-0.118 to 0.103] — Statistical data for IC
Statistical Analysis 7: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean difference of RV = -0.229, 95% CI 2-sided [-0.355 to -0.103] — Statistical data for RV
Statistical Analysis 8: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean difference of RV = -0.189, 95% CI 2-sided [-0.314 to -0.064] — Statistical data for RV
Statistical Analysis 9: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; Mean difference of TLC = -0.101, 95% CI 2-sided [-0.204 to 0.002] — Statistical data for TLC
Statistical Analysis 10: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.044, Mixed Models Analysis; Mean difference of TLC = -0.105, 95% CI 2-sided [-0.206 to -0.003] — Statistical data for TLC
Statistical Analysis 11: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg QD; Test type: Superiority or Other; p = 0.085, Mixed Models Analysis; Mean difference of TGV = -0.092, 95% CI 2-sided [-0.197 to 0.013] — Statistical data for TGV
Statistical Analysis 12: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.083, Mixed Models Analysis; Mean difference of TGV = -0.091, 95% CI 2-sided [-0.195 to 0.012] — Statistical data for TGV

10. Secondary Outcome: Post-dose FEV1/FVC Ratio (Measured at Trough) at Day 28 of Each Treatment Period
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FVC is defined as the amount of air that can forcibly be blown out after a full inspiration. FEV1 and FVC data was obtained by spirometry measurements.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population
Measure: Least Squares Mean (Standard Error); unit: Ratio of FEV1/FVC
Groups:
- Tio 18 µg BID: Participants received Tio 18 µg QD (morning) via a HandiHaler inhaler plus Ado matching placebo BID (morning and evening) via dry powder inhaler, in one of the three treatment periods. Each treatment period consisted of 4 weeks and separated by a 2-week washout period. Participants were provided with a salbutamol inhaler to be used as relief medication throughout the study.
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg BID | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
Ratio of FEV1/FVC | 0.500 (0.0052) | 0.472 (0.0052) | 0.492 (0.0052)
Statistical Analysis 1: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Tio 18 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; FEV1/FVC ratio = 0.027, 95% CI 2-sided [0.014 to 0.041] — Statistical data for FEV1/FVC ratio
Statistical Analysis 2: Comparison: Ado 50/250 µg BID+Tio 18 µg QD vs Ado 50/250 µg BID; Test type: Superiority or Other; p = 0.223, Mixed Models Analysis; FEV1/FVC ratio = 0.008, 95% CI 2-sided [-0.005 to 0.021] — Statistical data for FEV1/FVC ratio

11. Secondary Outcome: Use of Rescue Medication (Number of Occasions Per 24-hour Period) as Recorded in the Daily Record Card at Day 28 of Each Treatment Period
Description: Participants were given daily record cards for daily completion during the run-in, washout and treatment periods. Each morning, participants recorded the number of occasions in the last 24 hours when they had used their rescue medication (salbutamol) for symptomatic relief of COPD symptoms.
Time Frame: Day 28 of each treatment period (up to 35 days)
Population: mITT Population. Only those participants available who used rescue medication at the specified periods were analyzed (represented by n=X, X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Number of occasions
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Number analyzed (Participants) | 50 | 50 | 50
Number of occasions
  Treatment, n=20, 18, 17 | 0.2 (0.62) | 0.3 (0.82) | 0.2 (0.55)
  Washout, n=15, 15, 11 | 0.4 (0.81) | 0.5 (1.24) | 0.4 (1.01)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of administration of the study drug until follow-up contact (up to Week 18).
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants randomized to treatment, who had taken at least one dose of study medication.
Arm/Group | Ado 50/250 µg BID+Tio 18 µg QD | Tio 18 µg QD | Ado 50/250 µg BID
Serious Adverse Events (participants affected / at risk) | 2/52 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 15/52 | 8/51 | 11/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ado 50/250 µg BID+Tio 18 µg QD (N=52) | Tio 18 µg QD (N=51) | Ado 50/250 µg BID (N=51)
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ado 50/250 µg BID+Tio 18 µg QD (N=52) | Tio 18 µg QD (N=51) | Ado 50/250 µg BID (N=51)
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1
Pericoronitis (Infections and infestations) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.